CLINICAL TRIAL: NCT06100055
Title: The ReVo Study (REctal Irrigation VOlume Study - 'Low Versus High Volume Irrigation - Optimising Rectal Irrigation Volume in Evacuatory Dysfunction'; A Randomised Controlled Trial)
Brief Title: The ReVo Study: Low-volume vs High-volume Rectal Irrigation
Acronym: ReVo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 324658; 324658 (Other: IRAS)
Record Dates: First submitted 2023-10-10; First posted 2023-10-25 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Constipation - Functional; Constipation; Constipation by Outlet Obstruction; Defecation Disorder
Keywords: chronic constipation; rectal irrigation; evacuation disorders; low-volume rectal irrigation; high-volume rectal irrigation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: This is a superiority trial with parallel group design where each participant will receive only one of the two types of intervention (rectal irrigation).
Who Masked: Outcomes Assessor
Masking Description: Participants and clinicians will be aware of treatment allocations. The need to collect data on frequency and volume of irrigation, as well as reasons for discontinuing means that assessor blinding is not possible with respect to these outcomes. However, the statistician involved in the analysis will only receive coded data and therefore will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-volume rectal irrigation (Active Comparator): This system consists of a small reservoir attached to a cone. Depending on the manufacturer, the reservoir can hold approximately between 110ml and 300ml of water. This reservoir is squeezed to inject water into the rectum. The regime will be such that participants will be asked to use rectal irrigation daily for two weeks. They will be restricted to not use rectal irrigation for more than once in a day. Every day they can use up to 300ml for irrigation. After two weeks participants can then adjust the number of irrigation days per week as well as volume used for irrigation but not exceeding irrigation therapy more than once a day and not more than 300ml per irrigation. Volume and frequency of rectal irrigation will be recorded by participant in participant journal. This will be used to check their compliance and average weekly irrigation sessions and volume used for satisfactory outcome.
  Interventions: Device: Rectal Irrigation
- High-volume rectal irrigation (Active Comparator): The high-volume irrigation system consists of an irrigation bag connected to a tube. The water flows into the rectum, either by gravity or by using a pump. Some systems use balloon to hold the device in place during irrigation; others require the user to hold it in place. The mechanism of action is the same for all systems. Participants will start irrigation with 300ml and increase this by 100ml every 2 days until satisfactory defaecation is achieved, or the procedure becomes uncomfortable, up to a maximum of 1500ml. Initial frequency of irrigation is the same as for low-volume irrigation: i.e. once daily for two weeks followed by participant adjustment of number of irrigation days per week as well as volume used for irrigation but no more than 1500ml a day. Participants will be restricted to using high-volume irrigation to not more than once a day.
  Interventions: Device: Rectal Irrigation

INTERVENTIONS:
Device: Rectal Irrigation — Rectal irrigation is the introduction of warm tap water through the anal canal into the rectum to initiate defaecation.
  Two alternative irrigation systems based on volume delivered exist: low-volume irrigation system depending on the manufacturer delivers approximately between 110ml to 300ml per irrigation and high-volume irrigation system delivers between 300ml to 1500ml per irrigation.
  Other Names: trans-anal irrigation

SUMMARY:
Rectal irrigation, which is the introduction of warm tap water through the anal canal into the rectum to initiate defaecation, is recommended to be considered in patients with chronic constipation, which is refractory to conservative measures such as lifestyle modification, laxatives, nurse-led bowel retraining programmes which focuses on bio-feedback as well as psychosocial support.

Two systems of rectal irrigation are available based on volume delivered, low and high volume. It is unknown if one type of irrigation is superior to the other and whether one type has better outcomes in patients with a particular pathology.

Therefore, a comparison is required between the two types of irrigation to assess their acceptability as a therapy and response rates in patients with chronic constipation secondary to difficulty emptying rectum.

This trial/research aims to compare low-volume rectal irrigation with high-volume rectal irrigation in patients with chronic constipation secondary to disorders of difficulty emptying rectum.

The main questions it aims to answer are:

* if one type of rectal irrigation is superior to the other
* whether one type of rectal irrigation has better outcomes in patients with a particular pathology on pelvic floor ultrasound
* assess the acceptability and response rates to rectal irrigation.

Participants upon recruitment will be allocated to either low-volume rectal irrigation or high volume rectal irrigation groups. This will purely be by chance where the possibility of being in either of the groups will be 50%. They will then undergo a baseline assessment with four quality-of-life questionnaires and clinical examination. Following this a pelvic floor ultrasound will be performed to assess the cause of their symptoms. Lastly they will be provided training on using rectal irrigation (the type they have been assigned to). They will then be asked to commence irrigation at home from the next day.

Participants will continue to use irrigation for three months and then have a three-monthly follow-up where the quality of life questionnaires will be filled again. This data will then be used to assess any improvement in symptoms after using rectal irrigation. After three months of using rectal irrigation, participation in the trial will come to and end.

DETAILED DESCRIPTION:
Rectal irrigation(RI) is introducing warm tap water through the anal canal into the rectum to initiate defaecation. It is recommended that rectal irrigation be considered in patients with evacuation disorders refractory to conservative measures and bio-feedback before performing surgery.

RI is provided either as low-volume(LV) or high-volume(HV). It is unknown if one type of RI is superior to the other and whether one type of RI has better outcomes in patients with a particular pathology.

This randomised controlled trial aims to compare outcomes between two types of RI (LV and HV) and assess efficacy and acceptability of RI as a therapy in patients with Chronic constipation (CC) secondary to evacuation disorders (ED).

Primary Objective To compare the impact of LV RI versus HV RI, upon disease-specific quality of life at three months in patients with CC secondary to ED.

Secondary Objectives

* Improvement in participants' symptoms from RI by measuring symptoms severity score at three months.
* To identify if subgroup of participants with anatomical or pathophysiological variant of ED identified on integrated total pelvic floor ultrasound (TPFUS) will have different outcome from using RI
* Compliance to allocated type of RI and reasons for discontinuation.

Visit 0 (V0): Potentially eligible participants will be identified by the Co-investigator(TG) from Telephone triage assessment clinic, bio-feedback clinic(BFB) and Multi-Disciplinary Meeting in PFU at St. Thomas' Hospital. TG will introduce the research to eligible participants by contacting via telephone or during BFB.

Eligible participants will be provided with an information pack with invitation letter, participant information sheet (PIS) and two consent forms with a return label to post one of the consent forms back for record. PIS will have all details and explanation of the aims, methods, anticipated benefits and possible risks of RI. It will also have contact details of the Principle Investigator (PI) and the TG should eligible participants have any questions regarding the research trial before participating or to escalate concerns during participation. Participants will have at least 48 hours to consider participation.

Telephone Appointment (TA): This will scheduled at least 48 hours after the eligible participant has received the information pack. TG will contact the eligible participant to discuss the trial in detail and answer any queries. After discussion, if eligible participant is happy to participate, both consent forms will be signed. Participants will then be asked to return one consent form to the department for record (return label provided). There is no obligation for eligible participants to give reasons for non-participation.

Participants during the trial can withdraw anytime without giving reasons and return to routine care. However, data collected up to that point will be used to analyse current research as per PIS and consent form.

After consent, a participant journal (PJ) will be posted with instructions to fill it in. PJ will record all participants' medications and visits to healthcare professionals for constipation in the past three months. It will also record bowel frequency two weeks before participants' first face-to-face appointment.

Visit 1, Face-to-face (V1F): Baseline assessment, randomisation, TPFUS and training in RI Participants will have medical history taken and undergo a physical examination of their back passage and vagina (female participants). Participants will be asked to hand over PJ filled at home and fill in four questionnaires which will help investigators assess impact of constipation on participants' daily routine. These are PAC-QOL, PAC-SYM, ICIQ-B and ODS-S as described in outcome measures.

Participants will be randomly assigned 1:1 into two groups; LV RI and HV RI. Investigators will use online software (Clinical trial randomisation tool by National Cancer Institute) for randomisation. Both LV and HV irrigation will be given a code by TG. PI will perform randomisation and will perform allocation concealment using sealed envelopes.

Participants will undergo TPFUS which is routinely performed on all our patients. It uses inaudible sound waves to provide real-time static and dynamic multi-compartmental pelvic floor assessment of anatomical and functional aspects.

The RI systems used in our unit are commercially available on prescription in National Health Service (NHS) practice. Participants will receive training on using RI system from our Nurse Specialist and will be provided equipment to commence RI at home from the next day. Participants will be shown how to record the frequency and volume of RI in the PJ and record any side effects, such as pain, bleeding, etc.

Participants will be contacted via telephone one week later to check for any issues. If necessary, investigators will arrange another training.

Visit 2- face to face (V2F): This appointment will be three months after starting RI where participants will fill in outcome questionnaires as in previous visit and PJ will be collected. This will end participation in the research trial and participants will return to routine care in our department.

During 3-month follow-up, participants may be withdrawn from the trial if become lost to follow-up after at least three failed attempts by TG to make contact via at least two different methods (e.g., telephone, email and letter), choose to withdraw and do not wish to participate in follow-up data collection or lose capacity.

The interventions (LV and HV RI) proposed are those already being offered to patients with CC secondary to ED in the Pelvic Floor Unit(PFU), St. Thomas' Hospital and many specialist centres globally. All interventions pose acceptable risks. TPFUS has been performed routinely in most specialist centres and is considered safe. RI has proven to be a low-risk intervention and has been widely used for a variety of ED. Serious adverse events (SAE) are rare, with one study reporting two non-fatal bowel perforations out of approximately 110,000 irrigation therapy. Other possible side effects include rectal pain, bleeding, painful haemorrhoids and anal fissure. A recent study reported an overall adverse event (AE) rate of 22% with all minor and reversible events considered.

This trial is categorised as Type A i.e. no higher than the risk of standard medical care.

Any AE or SAE reported by participant will be reported to the sponsor and Ethical committee by the PI. The PI may take urgent safety measures to ensure the safety and protection of the participants. The PI will send the Annual Progress Report to the sponsor and Ethical committee.

If the PI determines that, is it within the best interests of the participants to terminate the study, written notification will be given to the sponsor following which participants will be returned to the routine NHS care.

The research team in the PFU will be meeting every two weeks. A trial risk assessment will be conducted in collaboration with the PI and an appropriate trial monitoring and auditing plan will be produced. This will be authorised by the sponsor.

PAC-QOL comprises of 28 questions scored 0-4. Average score of the non-missing questions is calculated by total score divided by number of questions responded, is taken as participant score out of 4. Considering improvement in score of 10% as clinically relevant, we calculated sample size keeping level of significance as 5%, power as 90% and standard deviation of 0.8 in low-volume RI and 0.7 in high-volume RI groups as reported by Emmett CC et al. Adjusting for loss to follow up of 10%, we will need 83 participants in each group. However, should there be a greater than 10% dropout rate which we do not feel will be the case, we will then recruit more participants to be able to analyse with a significance of 5% and power of 90%.

Primary outcome Investigators plan to conduct intention to treat analysis to compare the two types of RI at the end of 3 months. Difference in improvement in PAC-QOL score will be tested using paired sample t-test. Results will be reported as means along with standard deviations of difference in pre and post rectal irrigation for both groups and the mean difference of two interventions along with 95% confidence interval with p-value less than 0.05 will be taken as statistically significant.

Secondary outcomes Investigators plan to conduct stratified analysis based upon findings on TPFUS (anatomical vs functional causes of CC secondary to evacuation disorders). Compliance to RI will be shown via proportion of participants using it at the end of 3 months. Adverse effects from RI will be presented as frequencies. Appropriate regression models will be developed to determine the influence of pre-treatment characteristics on the success of RI in all sub-groups. Analysis will be performed using Statistical Package for the Social Sciences which is an online software platform where P < 0.05 will be taken to indicate statistical significance.

Investigators plan to conduct interim analysis at half the required sample size. At this point, the efficacy outcome will be evaluated and if the difference between two types of RI is statistically significant enough to reach p-value of < 0.01 then that would be considered as sufficient evidence to establish the superiority of one irrigation system over another and continuing the trial further would not be justified.

In the event of a required protocol amendment, details will be submitted to the sponsor for authorisation.

Data Protection: Upon recruitment, identifiable participant data (IPD) will be collected on paper (CRF) to contact participants. CRF will be stored in locked cabinets while electronic data in a password protected file(PPF) on Microsoft access (MA). Only PI and TG will have access to IPD.

TG will generate and assign a unique trial registration code (UTRC) to each participant. Each participant's data will be collected and stored against the UTRC (pseudonymization). CRF will be kept in locked cabinets while electronic data will be recorded in PPF on MA. The participant's general practitioner will be informed of their participation after obtaining consent.

After data collection has ended, TG will create a copy of collected data without the UTRC in a PPF on Microsoft Access, thus completely anonymising data which will be emailed to the Statistician via encrypted email for analysis.

This study is sponsored by Guy's and St Thomas' NHS Foundation Trust (GSTFT) and indemnity is provided through NHS indemnity for clinical negligence. GSTFT is a member of the clinical Negligence Scheme for Trusts.

The project will be under PI and sponsor. The project will be overseen by PI and co-Investigators. The role of the PI will be to provide overall supervision of the study on behalf of the sponsor to ensure that research trial is conducted in accordance with the principles of Good Clinical Practice (GCP) relevant regulations.

A study launch meeting will be conducted. This will include training in the trial protocol, data collection, randomisation and taking informed consent.

The participants will not be identifiable with regards to any future publications. After trial completion, the pseudonymized records will be kept for a further five years and archived with Iron Mountain. All IPD will also be archived for a period of five years in locked cabinets in the Pelvic Floor Unit at St. Thomas' Hospital, therefore no third party will have access to it. At the end of the five-year retention period, permission will be obtained in writing from the sponsor prior to destruction of this material.

Once results are available, they will first be presented in a departmental meeting, followed by submission of a summary to health research authority. A brief summary of the outcomes will be posted to the participants. Finally results will be submitted to scientific journals or presented at a conference not involving any IPD.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over 18 years who have self-reported problematic constipation secondary to evacuation disorders
* With symptom onset of more than 6 months
* Symptoms must meet American College of Gastroenterology definition of constipation which is symptoms including unsatisfactory defecation with either infrequent stools, difficulty in passing stool or both for at least previous 3 months (25)
* All should have tried and failed conservative management (laxatives, life-style modification and bio-feedback)
* Patients should also have ability and willingness to give informed consent.
* Patients or carer should be able to use rectal irrigation

Exclusion Criteria:

Patients with

* Major colorectal resection surgery, pelvic floor surgery to address defaecatory problems such as posterior vaginal repair, STARR, rectopexy and sacral nerve stimulation within last three months
* Pregnancy
* Active rectal bleeding
* Colorectal cancer
* Complicated diverticular disease or acute diverticulitis
* Anal or colorectal stenosis
* Inflammatory bowel disease
* Undergoing chemotherapy
* Ischemic colitis
* Used rectal irrigation in the past one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Patient Assessment of Constipation - Quality of Life questionnaire (PAC-QOL) | At baseline and after three months after using rectal irrigation
  PAC-QOL measures health related quality of life in patients with constipation. Lower score reflects better quality of life where it ranges from 0-112

SECONDARY OUTCOMES:
Patient Assessment of Constipation - Symptoms (PAC-SYM) | At baseline and after three months of using rectal irrigation
  PAC-SYM questionnaire assesses the severity of patient reported symptoms of constipation where score ranges from 0-48 where higher scores indicate more severe symptoms
Obstructed Defaecation Syndrome - Score (ODS-S) | At baseline and after three months of using rectal irrigation
  This questionnaire will be used to diagnose presence of Obstructive Defaecation Syndrome. A score >9 is diagnostic of ODS
International Consultation on Incontinence Questionnaire Anal Incontinence Symptoms and Quality of Life Module (ICIQ-B) | At baseline and after three months of using rectal irrigation
  Evaluates symptoms of anal incontinence and its impact on quality of life (QOL). Scores from 1-21 for bowel pattern, 0-28 for bowel control and 0-26 for impact on quality of life associated with anal incontinence symptoms where higher score is suggestive of worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Hainsworth, FRCS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No planned analysis other than current study

REFERENCES:
- [Background] Stewart WF, Liberman JN, Sandler RS, Woods MS, Stemhagen A, Chee E, Lipton RB, Farup CE. Epidemiology of constipation (EPOC) study in the United States: relation of clinical subtypes to sociodemographic features. Am J Gastroenterol. 1999 Dec;94(12):3530-40. doi: 10.1111/j.1572-0241.1999.01642.x. PMID 10606315
- [Background] Sonnenberg A, Koch TR. Epidemiology of constipation in the United States. Dis Colon Rectum. 1989 Jan;32(1):1-8. doi: 10.1007/BF02554713. PMID 2910654
- [Background] van den Berg MM, Benninga MA, Di Lorenzo C. Epidemiology of childhood constipation: a systematic review. Am J Gastroenterol. 2006 Oct;101(10):2401-9. doi: 10.1111/j.1572-0241.2006.00771.x. PMID 17032205
- [Background] Probert CS, Emmett PM, Heaton KW. Some determinants of whole-gut transit time: a population-based study. QJM. 1995 May;88(5):311-5. PMID 7796084
- [Background] Cook IJ, Talley NJ, Benninga MA, Rao SS, Scott SM. Chronic constipation: overview and challenges. Neurogastroenterol Motil. 2009 Dec;21 Suppl 2:1-8. doi: 10.1111/j.1365-2982.2009.01399.x. PMID 19824933
- [Background] Wald A, Scarpignato C, Mueller-Lissner S, Kamm MA, Hinkel U, Helfrich I, Schuijt C, Mandel KG. A multinational survey of prevalence and patterns of laxative use among adults with self-defined constipation. Aliment Pharmacol Ther. 2008 Oct 1;28(7):917-30. doi: 10.1111/j.1365-2036.2008.03806.x. Epub 2008 Jul 17. PMID 18644012
- [Background] Irvine EJ, Ferrazzi S, Pare P, Thompson WG, Rance L. Health-related quality of life in functional GI disorders: focus on constipation and resource utilization. Am J Gastroenterol. 2002 Aug;97(8):1986-93. doi: 10.1111/j.1572-0241.2002.05843.x. PMID 12190165
- [Background] Knowles CH, Grossi U, Horrocks EJ, Pares D, Vollebregt PF, Chapman M, Brown SR, Mercer-Jones M, Williams AB, Hooper RJ, Stevens N, Mason J; NIHR CapaCiTY working group; Pelvic floor Society. Surgery for constipation: systematic review and clinical guidance: Paper 1: Introduction & Methods. Colorectal Dis. 2017 Sep;19 Suppl 3:5-16. doi: 10.1111/codi.13774. PMID 28960925
- [Background] Knowles CH, Dinning PG, Pescatori M, Rintala R, Rosen H. Surgical management of constipation. Neurogastroenterol Motil. 2009 Dec;21 Suppl 2:62-71. doi: 10.1111/j.1365-2982.2009.01405.x. PMID 19824939
- [Background] Knowles CH, Scott M, Lunniss PJ. Outcome of colectomy for slow transit constipation. Ann Surg. 1999 Nov;230(5):627-38. doi: 10.1097/00000658-199911000-00004. PMID 10561086
- [Background] Shandling B, Gilmour RF. The enema continence catheter in spina bifida: successful bowel management. J Pediatr Surg. 1987 Mar;22(3):271-3. doi: 10.1016/s0022-3468(87)80345-7. PMID 3550032
- [Background] Briel JW, Schouten WR, Vlot EA, Smits S, van Kessel I. Clinical value of colonic irrigation in patients with continence disturbances. Dis Colon Rectum. 1997 Jul;40(7):802-5. doi: 10.1007/BF02055436. PMID 9221856
- [Background] Christensen P, Krogh K. Transanal irrigation for disordered defecation: a systematic review. Scand J Gastroenterol. 2010 May;45(5):517-27. doi: 10.3109/00365520903583855. PMID 20199336
- [Background] Gardiner A, Marshall J, Duthie G. Rectal irrigation for relief of functional bowel disorders. Nurs Stand. 2004 Nov 10-16;19(9):39-42. doi: 10.7748/ns2004.11.19.9.39.c3755. PMID 15574053
- [Background] Crawshaw AP, Pigott L, Potter MA, Bartolo DC. A retrospective evaluation of rectal irrigation in the treatment of disorders of faecal continence. Colorectal Dis. 2004 May;6(3):185-90. doi: 10.1111/j.1463-1318.2004.00584.x. PMID 15109384
- [Background] Koch SM, Melenhorst J, van Gemert WG, Baeten CG. Prospective study of colonic irrigation for the treatment of defaecation disorders. Br J Surg. 2008 Oct;95(10):1273-9. doi: 10.1002/bjs.6232. PMID 18720454
- [Background] Emmett C, Close H, Mason J, Taheri S, Stevens N, Eldridge S, Norton C, Knowles C, Yiannakou Y. Low-volume versus high-volume initiated trans-anal irrigation therapy in adults with chronic constipation: study protocol for a randomised controlled trial. Trials. 2017 Mar 31;18(1):151. doi: 10.1186/s13063-017-1882-y. PMID 28359279
- [Background] Hainsworth AJ, De Robles MS, Ferrari L, Solanki D, Williams AB, Schizas A. Total pelvic floor ultrasound can reliably predict long-term treatment outcomes for patients with pelvic floor defaecatory dysfunction. Neurourol Urodyn. 2023 Jan;42(1):90-97. doi: 10.1002/nau.25051. Epub 2022 Sep 24. PMID 36153653
- [Background] Dietz HP. Pelvic Floor Ultrasound: A Review. Clin Obstet Gynecol. 2017 Mar;60(1):58-81. doi: 10.1097/GRF.0000000000000264. PMID 28005595
- [Background] Camilleri M, Kerstens R, Rykx A, Vandeplassche L. A placebo-controlled trial of prucalopride for severe chronic constipation. N Engl J Med. 2008 May 29;358(22):2344-54. doi: 10.1056/NEJMoa0800670. PMID 18509121
- [Background] Christensen P, Krogh K, Buntzen S, Payandeh F, Laurberg S. Long-term outcome and safety of transanal irrigation for constipation and fecal incontinence. Dis Colon Rectum. 2009 Feb;52(2):286-92. doi: 10.1007/DCR.0b013e3181979341. PMID 19279425
- [Background] American College of Gastroenterology Chronic Constipation Task Force. An evidence-based approach to the management of chronic constipation in North America. Am J Gastroenterol. 2005;100 Suppl 1:S1-4. doi: 10.1111/j.1572-0241.2005.50613_1.x. No abstract available. PMID 16008640
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Background] Renzi A, Brillantino A, Di Sarno G, d'Aniello F. Five-item score for obstructed defecation syndrome: study of validation. Surg Innov. 2013 Apr;20(2):119-25. doi: 10.1177/1553350612446354. Epub 2012 May 17. PMID 22599920
- [Background] Cotterill N, Norton C, Avery KN, Abrams P, Donovan JL. Psychometric evaluation of a new patient-completed questionnaire for evaluating anal incontinence symptoms and impact on quality of life: the ICIQ-B. Dis Colon Rectum. 2011 Oct;54(10):1235-50. doi: 10.1097/DCR.0b013e3182272128. PMID 21904138